CLINICAL TRIAL: NCT03316365
Title: Long-term Training Effects of Rhythmic Auditory Stimulation on Gait in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Poudre Valley Health System Fort Collins CO (Unknown); Colorado State University (Other)
Responsible Party: Principal Investigator, Michael H. Thaut, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-785
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Continuous Rhythmic Auditory Stimulation; Intermittent Rhythmic Auditory Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Home training instructions were provided by a certified physical therapist and board-certified neurologic music therapist blinded to treatment allocation of the subjects.
  The TUG and the BBS were administered by an experienced physical therapist blinded to the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous RAS (Experimental): The experimental group (continuous treatment) trained daily with RAS for 24 weeks.
  Interventions: Other: Rhythmic Auditory Stimulation (RAS)
- Intermittent RAS (Active Comparator): The control group (intermittent treatment) trained with RAS for 8 weeks, discontinued training for 8 weeks, and resumed training with RAS for 8 weeks.
  Interventions: Other: Rhythmic Auditory Stimulation (RAS)

INTERVENTIONS:
Other: Rhythmic Auditory Stimulation (RAS) — The experimental group (continuous treatment) trained daily with Rhythmic Auditory Stimulation (RAS) for 24 weeks. The control group (intermittent treatment) trained with RAS for 8 weeks, discontinued training for 8 weeks, and resumed training with RAS for 8 weeks. During treatment subjects walked for 30 minutes in a home-based environment with metronome-click embedded music downloaded to an MP3 player and listened to either free-field or via headphones. For the first 8 weeks subjects had 3 metronome rates available to choose from: 100, 105, and 110% of internal usual cadence. During the second 8 weeks available rates were 105, 110 and 115%; and during the last 8 weeks 110, 115, 120%. The control group started their last training segment at 105, 110, and 115%, but could request a change to the faster rates if comfortable.
  Other Names: Neurologic Music Therapy

SUMMARY:
Falls are common among patients with Parkinson's Disease (PD) and are the biggest contributors to loss of independent living, long-term institutionalization, and increased mortality.

The purpose of this study was to explore whether an at-home based Rhythmic Auditory Stimulation (RAS) gait training program will decrease the number of falls in persons with PD with a history of falling. We also evaluated changes in clinical and kinematic parameters used to assess fall risk in this population.

Sixty participants diagnosed with idiopathic PD with at least 2 falls in the past 12 months, were randomly allocated into two groups. The experimental group trained daily with RAS for 24 weeks. The control group also trained daily with RAS, but discontinued training between weeks 8 and 16. During treatment patients walked for 30 minutes in a home based environment with metronome-click embedded music. Changes in clinical and kinematic parameters were assessed at baseline, weeks 8, 16, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr (HY) stage III or IV
* At least 2 falls in the past 12 months
* Stable antiparkinsonian medication regime
* Ability to ambulate independently for at least 50 m.

Exclusion Criteria:

* Other neurological or orthopedic conditions
* Medically diagnosed hearing loss
* Dementia (Mini Mental Status Exam score < 24).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Fall Index | Change of the number of fall incidents and severity from baseline assessed by the Fall Index 8 weeks, 16 weeks, and 24 weeks.
  The Fall Index was computed based on self-reports by subjects or caregivers and classified as 1 (incomplete fall, lost balance but stabilized by another person or object), 2 (complete fall, no injuries) or 3 (complete fall, injury, medical attention required). A complete fall was defined as unintentionally coming to the ground with any body part above ankle. Higher Fall Index values indicate higher incidence of falls.

SECONDARY OUTCOMES:
Falls Efficacy Scale (FES) | Change in level of concern about falling from baseline assessed by Fear of the Falling Questionnaire/Short FES-1 at 8 weeks, 16 weeks, and 24 weeks.
  Falls Efficacy Scale (FES) (Tinetti et al 1990) is a 10-item scale to assess fear of falling in older persons. Individuals are asked to rate, on a 10-point scale with zero corresponding to not at all and 10 to completely, how confident he or she felt in performing 10 activities. The scores are added up to calculate a total score that ranges from 0 to 100. Higher scores indicate more confidence/less fear.
Berg Balance Scale (BBS) | Change in balance from baseline assessed by Berg Balance Scale at 8 weeks, 16 weeks, and 24 weeks.
  It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function, and the final measure is the sum of all of the scores.
Timed Up and Go (TUG) | Change in balance and function from baseline assessed by Timed Up and Go at 8 weeks, 16 weeks, and 24 weeks.
  Measure of function (rise from a chair, walk three meters, turn around, walk back to the chair, and sit down) with correlates to balance and fall risk. A faster time indicates a better functional performance.
Gait | Change in gait from baseline at 8 weeks, 16 weeks, and 24 weeks.
  Assessment of gait parameters (velocity, stride length, cadence, ankle dorsiflexion) with a computerized stride analyzer system (B&L Engineering).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thaut, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to external researchers.